CLINICAL TRIAL: NCT01333072
Title: Biomarkers in Autism of Aripiprazole and Risperidone Treatment
Brief Title: Biomarkers in Autism of Aripiprazole and Risperidone Treatment (BAART)
Acronym: BAART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R01HD062550-01A1 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2011-04-11 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Autistic Disorder
Keywords: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone (Active Comparator): Atypical antipsychotic
  Interventions: Drug: Risperidone
- Aripiprazole (Active Comparator): Atypical antipsychotic
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — The starting dosage will be 2.0 mg/day. The dosage will be allowed to increase to 5.0 mg/day on day 4 and can be increased thereafter as judged clinically appropriate until the maximum dosage of 15 mg/day. The dosage will only be increased in 5.0 mg intervals. No dosage adjustments will be allowed for either drug after 4 weeks.
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Risperidone — Children weighing 20-45 kg will receive an initial dose of 0.5 mg daily that will be increased to twice daily on day 4 (morning and bedtime). The dosage will be gradually increased in 0.5 mg increments to a maximum dose of 2.5 mg per day (1.0 mg in the morning and 1.5 mg at bedtime) by the fourth treatment week. A slightly accelerated dosage will be allowed for children who weigh more than 45 kg for a maximum dosage of 3.5 mg /day (McCracken et al 2002).
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
The Biomarkers in autism of aripiprazole and risperidone treatment (BAART) project will provide evidence-based guidance in the selection and monitoring of drug treatment of autism. BAART involves 3 academic centers across South Carolina. Although the FDA has approved use of the antipsychotic drug risperidone for irritability associated with autistic disorder, a moderate response rate in pivotal clinical trials and concerns over tolerability and weight gain can force clinicians to select alternative drug treatments for which evidence-based support is sparse.

DETAILED DESCRIPTION:
The Biomarkers in autism of aripiprazole and risperidone treatment (BAART) project will provide evidence-based guidance in the selection and monitoring of drug treatment of autism. BAART involves 3 academic centers across South Carolina with expertise in phenotyping patients with autistic spectrum disorders, assessing patient response in clinical trials, and expertise in pharmacogenomic research. Although the FDA has approved use of the antipsychotic drugs risperidone and aripiprazole for irritability associated with autistic disorder, a moderate response rate in pivotal clinical trials and concerns over tolerability and weight gain can force clinicians to select alternative drug treatments for which evidence-based support is sparse. BAART will assess predictors of efficacy, tolerability, and safety in 200 children 6-17 years old with autistic disorder (AD) during a double-blind, randomized 10 week treatment period with either risperidone or aripiprazole. Responders who complete the study may continue with medication treatment for three months. Factors considered will include 1) psychiatric history; 2) symptom response; 3) psychosocial support; 4) measures of tolerability; 5) serum prolactin and brain-derived neurotrophic factor concentration; and 5) a variety of single nucleotide polymorphisms related to target genes for drug disposition and transport, response, and tolerability. The BAART project will result in evidence-based guidelines for selection and monitoring of drug treatment of children and adolescents with AD.

ELIGIBILITY:
Inclusion Criteria

* Aged 6 to 17 years and weight of at least 15 kg
* Meet DSM-IV criteria for of AD, established by chart review, clinical judgment and the Autism Diagnostic Interview- Revised (ADI-R) criteria
* Clinical Global Impressions Severity (CGI-S) score of >4 (moderately ill)
* ABC Irritability subscale score of >18
* Mental age of at least 18 months
* If female and sexually active, must agree to an acceptable method of birth control during the trial
* Medication free or adequate washout period (2-4 weeks prior to enrollment) of psychoactive drugs (anticonvulsants permitted for seizure management if dosage is stable for 4 weeks)
* Parent/guardian able to read and provide informed consent.

Exclusion Criteria

* Psychiatric disorder that is effectively managed by psychoactive medication (e.g. ADHD, MDD)
* Prior diagnosis or evidence of genetic or other disorder that may interfere with assessments (e.g. Fragile X syndrome, Fetal alcohol syndrome, history of very low birth weight) assessed by personal and family history, dysmorphology, and clinical judgment.
* Prior use of risperidone or aripiprazole for more than 2 weeks
* Seizure during the past 6 months
* History or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments during the trial including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, hematologic or immunologic disease as determined by the clinical judgment of the investigator
* Current suicidal or homicidal risk
* Positive urine pregnancy test at baseline
* Dependent on other substances, with the exception of nicotine or caffeine

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2011-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Lindsay DeVane, Pharm.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] DeVane CL, Charles JM, Abramson RK, Williams JE, Carpenter LA, Raven S, Gwynette F, Stuck CA, Geesey ME, Bradley C, Donovan JL, Hall AG, Sherk ST, Powers NR, Spratt E, Kinsman A, Kruesi MJ, Bragg JE Jr. Pharmacotherapy of Autism Spectrum Disorder: Results from the Randomized BAART Clinical Trial. Pharmacotherapy. 2019 Jun;39(6):626-635. doi: 10.1002/phar.2271. Epub 2019 May 29. PMID 31063671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 participants were enrolled but 19 dropped from the study due to placebo response (16), parent withdrew child (2) and physician withdrew 1 subject. This left 61 subjects for randomization, as specified
Groups:
- Risperidone: Atypical antipsychotic
  Risperidone: Children weighing 20-45 kg will receive an initial dose of 0.5 mg daily that will be increased to twice daily on day 4 (morning and bedtime). The dosage will be gradually increased in 0.5 mg increments to a maximum dose of 2.5 mg per day (1.0 mg in the morning and 1.5 mg at bedtime) by the fourth treatment week. A slightly accelerated dosage will be allowed for children who weigh more than 45 kg for a maximum dosage of 3.5 mg /day.
Period: Overall Study
Arm/Group | Risperidone | Aripiprazole
Started | 30 | 31
Completed | 24 | 27
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 2 | 4
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone | Aripiprazole | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Median (Full Range); unit: years] | 8.3 [6.3 to 17.5] | 8.5 [6.0 to 15.1] | 8.4 [6.0 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 23 | 25 | 48
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Irritability Subscale of the Larger ABC (Abberent Behavior Checklist) That Occur From Baseline to 10 Weeks
Description: Multi-center, blinded clinical trial to evaluate biomarkers as predictors of efficacy and safety in children with autistic disorder to risperidone, an atypical antipsychotic drug and aripiprazole, an antipsychotic having a unique clinical and receptor-binding profile.
  The major outcome measure was the score on the Irritability subscale of the Aberrant Behavior Checklist (ABC-I) . The ABC has 58 items describing some aspect of behavior and the Irritability sub-scale has 15 items, each completed by a parent or caregiver under the supervision of an investigator. Scores on each item range from 0 = no problem and 3 = severe problem (range of total scores 0 to 45). A fall in scores indicates behavioral improvement.
Time Frame: baseline to 10 weeks
Population: Score on Aberrant Behavior Checklist (ABC) scale for Irritability
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone | Aripiprazole
Number analyzed (Participants) | 24 | 27
units on a scale | 12.7 (3.0) | 14.1 (3.5)

ADVERSE EVENTS:
Arm/Group | Risperidone | Aripiprazole
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 23/30 | 19/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=30) | Aripiprazole (N=31)
sedation (Psychiatric disorders) | 2 | 7
weight gain (Metabolism and nutrition disorders) | 21 | 8
enuresis (Psychiatric disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No